CLINICAL TRIAL: NCT03589417
Title: Postural Stability, Balance and Fall Risk in Patients With Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Melih Zeren, Principal Investigator, Bezmialem Vakif University
Other Study IDs: bvumzeren02
Record Dates: First submitted 2018-07-05; First posted 2018-07-17 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessments with Biodex Balance System® — Postural Stability, limits of stability and fall risk tests will be applied with the Biodex Balance System®

SUMMARY:
Obstructive sleep apnea (OSA) is a clinical condition characterized by the repetitive obstruction of the upper airway during sleep, resulting in nocturnal hypoxaemia and fragmented sleep. Fragmented sleep leads to daytime sleepiness that causes alterations in reaction times and reflexes . Postural stability is an important function of the human body. It is shown that the sleep deprivation disturbs daytime postural stability and balance. Aim of this study is to examine the influence of OSA severity and daytime sleepiness on postural stability, balance and fall risk.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with recent diagnosis of OSA (AHI≥5)
* BMI of ≤35 kg/m2
* Being sedentary

Exclusion Criteria:

* Having OSA treatments (CPAP, oral devices, nasal surgery, tennis ball/positional therapy, diuretic),
* Having a disease that can affect balance (vestibular, neurological, orthopedic ...) performing regular exercise
* Morphological defect (facial malformation, etc.) which may cause sleep disorders
* Uncontrolled hypertension or arrhythmia
* History of smoking or alcoholism
* Orthopedic, neurological or musculoskeletal problems which impede exercising
* Pregnancy
* Uncompensated clinical conditions such as chronic obstructive pulmonary disease, interstitial lung disease, heart failure, or rheumatic and psychiatric diseases

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects aged between 30-65 years who are recently diagnosed with mild, moderate or severe OSA (AHI≥5) and not receiving any treatment yet will be included in the study.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
Postural Stability Test score | Baseline
  'Postural Stability Test' will be applied with Biodex Balance System®. Subjects will stand still on the platform and the displacement of the centre of gravity will be quantified for anterior-posterior (AP) and medial-lateral (ML) axes. Test provides three types of scores: overall stability index, anterior-posterior stability index and medial-lateral stability index. Higher scores indicate worse postural stability.
Limits of Stability Test score | Baseline
  'Limits of Stability Test' will be applied with Biodex Balance System®. Subjects will stand on the platform and lean in eight directions to control the cursor displayed on the screen and try to move the cursor inside the target circles. Test provides scores for all eight directions as well as an overall score. Higher scores indicate better performance (0= worst performance; 100= perfect performance)
Fall risk Test score | Baseline
  'Fall Risk Test' will be applied with Biodex Balance System®. Subjects will stand still on the platform which will gradually become more unstable for 20 seconds. Total displacement of the centre of gravity will be quantified. Test provides one score: Overall stability index. Higher score indicates higher risk of fall.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif Universitesi, Department of Physiotherapy and Rehabilitation, Istanbul, Eyup, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yilmaz Gokmen G, Gurses HN, Zeren M, Ozyilmaz S, Kansu A, Akkoyunlu ME. Postural stability and fall risk in patients with obstructive sleep apnea: a cross-sectional study. Sleep Breath. 2021 Dec;25(4):1961-1967. doi: 10.1007/s11325-021-02322-2. Epub 2021 Feb 20. PMID 33608798